CLINICAL TRIAL: NCT06104319
Title: A Phase 2a, Single Dose, Open-label, Dose Exploration Study to Assess the PK-PD Activity, Safety, and Tolerability of GSK4532990 in Adult. Participants With NASH or Suspected NASH
Brief Title: Dose Exploration Study of GSK4532990 in. Participants With NASH or Suspected NASH
Acronym: SKYLINE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 218675
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: GSK4532990; Non-alcoholic steatohepatitis (NASH); Non-alcoholic fatty liver disease (NAFLD); Suspected NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- GSK4532990 Dose 1 (Experimental): Participants will receive GSK4532990 Dose 1
  Interventions: Drug: GSK4532990
- GSK4532990 Dose 2 (Experimental): Participants will receive GSK4532990 Dose 2
  Interventions: Drug: GSK4532990
- GSK4532990 Dose 3 (Experimental): Participants will receive GSK4532990 Dose 3
  Interventions: Drug: GSK4532990
- GSK4532990 Dose 4 (Experimental): Participants will receive GSK4532990 Dose 4
  Interventions: Drug: GSK4532990

INTERVENTIONS:
Drug: GSK4532990 — GSK4532990 will be administered

SUMMARY:
The purpose of this study is to understand how the drug GSK4532990 is processed in the body (pharmacokinetics) and how it works in the liver (pharmacodynamics) as well as to ensure it is safe and well-tolerated. The total study duration for each participant will be approximately 24-36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 75 years of age.
* Participant must be capable of giving signed informed consent which includes compliance with the requirements and restrictions listed for the study.
* Participants who have proven diagnosis of NASH or suspected NASH based on defined study criteria.
* Participants must meet predefined stable use requirements of concomitant medications based on study criteria.

Exclusion Criteria:

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

* Cirrhosis or current unstable liver or biliary disease.
* Other causes of liver disease including, but not limited to, alcohol-related liver disease, autoimmune disorders.
* Known weight loss of ≥5% within 3 months prior to Screening.
* Weight reduction surgery or procedures within 2 years of Screening.
* Any contraindication to undergoing liver biopsy.
* Any contraindication to undergoing Magnetic Resonance Imaging or FibroScan®.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Predicted percent change from baseline in liver biopsy-derived HSD17B13 protein expression levels | Baseline (Day 1) and up to Week 28
Predicted percent change from baseline in liver biopsy-derived HSD17B13 mRNA expression levels | Baseline (Day 1) and up to Week 28

SECONDARY OUTCOMES:
Area under the concentration-time curve from time zero (pre-dose) to the last quantifiable concentration (AUC0-t) of GSK4532990 | Pre-dose (Day 1), 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 and 48 hours post dose
Maximum observed concentration (Cmax) of GSK4532990 | Pre-dose (Day 1), 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 and 48 hours post dose
Percent change from baseline in the. observed HSD17B13 protein expression. levels | Baseline and Weeks 8, 12, or 28 post-dose
Percent change from baseline in the. observed HSD17B13 mRNA expression. levels | Baseline and Weeks 8, 12, or 28 post-dose

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, Montclair, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Lakes, Florida
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, El Dorado, Kansas
  - GSK Investigational Site, Marrero, Louisiana
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/